CLINICAL TRIAL: NCT03885297
Title: Investigation of the Metabolic Effects of 3mg Liraglutide on Patients With Overweight or Obesity
Brief Title: 3mg Liraglutide for Overweight or Obesity
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Kingston University (Other); University of Warwick (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: GD410218; 250896 (Registry Identifier: IRAS ID number)
Record Dates: First submitted 2019-02-27; First posted 2019-03-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Overweight; Obesity; Infertility, Female
Keywords: obesity; metabolism; liraglutide; saxenda; metabolomics; miRNA; weight loss
MeSH Terms: conditions — Overweight; Obesity; Infertility, Female; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overweight/obese participants: Patients will be recruited prospectively from the weight management and Polycystic Ovary Syndrome (PCOS) clinics at University Hospitals Coventry and Warwickshire (UHCW) NHS Trust following discussion with their treating physician, who will also be a member of the research team and joint agreement on initiation of treatment with 3mg Liraglutide once daily as per clinical management plan. Patients will additionally receive standard NHS Tier 3 lifestyle advice and support for the duration of the study. Lifestyle modification aimed at weight loss will be delivered by a dietician or other trained health care professional within individual sessions for a period of 6 months. Finally, all patients will be able to withdraw from treatment and/or the study at any point without giving any explanation. This will have no impact in their clinical management.
  Interventions: Drug: Saxenda; Other: Lifestyle modification; Diagnostic Test: Metabolomics; Diagnostic Test: miRNA

INTERVENTIONS:
Drug: Saxenda — Obesity pharmacotherapy
Other: Lifestyle modification — Tier 3 NHS weight management
Diagnostic Test: Metabolomics — Small molecule intermediates and products of metabolism
Diagnostic Test: miRNA — Small non-coding RNA molecules

SUMMARY:
In this study investigators will investigate the beneficial metabolic sequelae of Liraglutide in patients with obesity or overweight; including changes in vital signs, anthropometric characteristics (weight, body mass index and body composition), biochemical parameters, metabolomics and micro-ribonucleotide acid (miRNA) molecules from blood tests. Liraglutide is a commercially available analogue of a gut hormone physiologically produced in our bowel in response to food, licenced for the treatment of overweight or obesity. Liraglutide will be offered to patients attending National Health System (NHS) or private clinics within indication and according to their agreed clinical management. Investigators aim to collect real-life information for this study along with planned clinical management from patients who agree to their treatment and to take part in our study. Patients will be able to withdraw from treatment and study at any time without giving any explanation.

If successful, this study will help us combine clinical, biochemical and molecular information which will allow us to gain deeper understanding on the mechanisms behind the beneficial metabolic effects of Liraglutide in overweight and obesity. Data generated from this study will hopefully help us acquire funding for a larger multicentre study; the results of which can have substantial impact on millions of people with overweight or obesity around the world.

DETAILED DESCRIPTION:
1) Obesity is a global pandemic with debilitating consequences. It affects both adults and children; however, the prevalence of overweight and obesity among children and adolescents aged 5-19 has risen dramatically from just 4% in 1975 to just over 18% in 2016, highlighting the seriousness of this problem. The rise has occurred similarly among both boys and girls: in 2016 18% of girls and 19% of boys were overweight. While just under 1% of children and adolescents aged 5-19 were obese in 1975, more 124 million children and adolescents (6% of girls and 8% of boys) were obese in 2016.

Obesity is a major risk factor for noncommunicable diseases such as:

1. Cardiovascular diseases (mainly heart disease and stroke), which were the leading cause of death in United States of America(USA);
2. Diabetes Mellitus
3. Musculoskeletal disorders (especially osteoarthritis - a highly disabling degenerative disease of the joints);
4. Some forms of malignancy (including endometrial, breast, ovarian, prostate, liver, gallbladder, kidney, and colon);
5. Infertility in both women and men. The risk for these noncommunicable diseases increases, with increases in Body Mass Index (BMI).

2) Liraglutide is a derivative of human incretin (metabolic hormone) glucagon-like peptide-1 (GLP-1) that is used as a long-acting glucagon-like peptide-1 receptor agonist, binding to the same receptors as does the endogenous metabolic hormone GLP-1 that stimulates insulin secretion. Liraglutide is licenced in USA and in European Union (EU), including United Kingdom (UK) for the management of Type 2 Diabetes Mellitus (T2DM) and Obesity or overweight when one or more metabolic co-morbidities are present.

Saxenda (3mg Liraglutide once daily) is an Food & Drug Administration (FDA)-approved, prescription injectable Glucagon Like Peptide-1 (GLP-1) receptor agonist that, when used with a low-calorie diet and increased physical activity, can reduce excess weight in patients who are overweight (BMI ≥27Kg/m2) and additionally have weight-related medical problems (such as high blood pressure, high cholesterol, or insulin resistance/pre-diabetes), or obesity (BMI: >30Kg/m2) to lose weight. Saxenda is licensed and available in the UK for the management of obesity and overweight.

3) Metabolomics is the scientific study of chemical processes involving metabolites, the small molecule intermediates and products of metabolism. Specifically, metabolomics is the "systematic study of the unique chemical fingerprints that specific cellular processes leave behind", the study of their small-molecule metabolite profiles. The metabolome represents the complete set of metabolites in a biological cell, tissue, organ or organism, which are the end products of cellular processes. This in emerging area of metabolic research and in this study, will provide insight into the mechanisms through which 3mg Liraglutide improves weight and other metabolic sequelae (i.e glucose and lipids homeostasis) in humans during treatment. To the extend of our knowledge, there is a very limited number of such studies; none of which reporting on the effects of 3mg Liraglutide. Our collaborator Professor Gyanendra Tripathi has kindly agreed to fund costs for metabolomics analysis of our human samples. Metabolomics analysis of human serum or plasma samples is going to be performed by applying Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS). UPLC-MS assay will provide untargeted study of water-soluble metabolites (HILIC LCMS) and untargeted study of lipid metabolites (C18 reversed phase LCMS). Analysis is going to be performed at School of Biosciences, University of Birmingham.

4) MicroRNA (abbreviated miRNA) is a small non-coding RNA molecule (containing about 22 nucleotides) found in plants, animals and some viruses, that functions in RNA silencing and post-transcriptional regulation of gene expression. While most miRNAs are located within the cell, some miRNAs, commonly known as circulating miRNAs or extracellular miRNAs, have also been found in extracellular environment, including various biological fluids and cell culture media. MiRNAs play crucial roles in the regulation of stem cell progenitors differentiating into adipocytes. Studies to determine what role pluripotent stem cells play in adipogenesis, were examined in the immortalized human bone marrow-derived stromal cell line hMSC-Tert20. Decreased expression of miRNA-155, miRNA-221, and miRNA-222, have been found during the adipogenic programming of both immortalized and primary human Mesenchymal Stem Cells (hMSCs), suggesting that they act as negative regulators of differentiation. Conversely, ectopic expression of the miRNAs 155,221, and 222 significantly inhibited adipogenesis and repressed induction of the master regulators Peroxisome proliferator-activated receptor gamma(PPARγ) and CCAAT/enhancer-binding protein alpha (CEBPA). This paves the way for possible genetic obesity treatments. Our goal is however to see if treatment with 3mg Liraglutide will influence circulating miRNA levels. To the extent of our knowledge there is currently no study reporting this.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants [age ≥18 y.o without upper age limit (to the discretion of the investigators)].
* Body mass index (BMI) ≥ 30 kg/m2 without coexisting comorbidities or BMI ≥27Kg/m2 with comorbidities like hypertension, hyperlipidaemia, prediabetes or obstructive sleep apnoea.
* Willing to comply with study requirements and able to give informed consent.

Exclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* History of chronic or acute pancreatitis
* Known active hepatitis or active liver disease
* Symptomatic gallstones or kidney stones, acute cholecystitis or history of duodenal inflammatory diseases including Crohn's Disease and Celiac Disease
* Persistent anaemia, defined as haemoglobin<10 g/dl
* Chronic or acute renal impairment (eGFR <30 ml/min/1.73m2)
* Active systemic infection (sepsis)
* Active malignancy within the last 5 years, including any form of thyroid cancer (including sporadic or familial medullary thyroid cancer) or personal, or family history of Multiple Endocrine Neoplasia type 2.
* Active illicit substance abuse or alcoholism
* Current pregnancy or breastfeeding at screening or 6 months previously
* Donated blood during the preceding 3 months or intention to do so before the end of the study.
* Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators don't anticipate any specific difficulties with recruitment for this study as overweight and obesity are very common conditions, and there are very few licensed medical options offering substantial weight loss. Liraglutide is one of them. Additionally, investigators don't see any specific difficulties in managing this study as it will be " part and parcel" of our patients' routine clinical visits. Liraglutide is going to be offered to our patients as per clinical need and the decision to treat them with liraglutide is going to be made before their potential participation in our study. Patients therefore are not going to be receiving treatment because of their participation in our study.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Weight changes related to treatment | 6 months
  Weight reduction in kilograms from baseline while on treatment with 3mg Liraglutide once daily in patients with overweight (BMI: ≥27Kg/m2) or obesity (BMI: ≥30Kg/m2) with regards to:

SECONDARY OUTCOMES:
Changes in fat and lean mass while on treatment | 6 months
  Fat and lean mass changes in percentages from baseline using air displacement plethysmography and bioelectrical impedance techniques while on treatment with 3mg Liraglutide once daily for overweight and obesity
Changes in an untargeted study of water-soluble metabolites (HILIC LCMS) while on treatment | 6 months
  Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS) will be performed to measure plasma changes of water-soluble metabolites (HILIC LCMS).
Changes in an untargeted study of lipid metabolites (C18 reversed phase LCMS) while on treatment | 6 months
  Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS) will be performed to measure plasma changes of lipid metabolites (C18 reversed phase LCMS)
Changes in the expression of miRNA-155 while on treatment. | 6 months
  Decreased expression of miRNA-155 has been found during the adipogenic programming of both immortalized and primary hMSCs, suggesting that it acts as negative regulators of fat cell differentiation. We will measure this in plasma.
Changes in the expression of miRNA-221 while on treatment. | 6 months
  Decreased expression of miRNA-221 has been found during the adipogenic programming of both immortalized and primary hMSCs, suggesting that it acts as negative regulators of fat cell differentiation. We will measure this in plasma.
Changes in the expression of miRNA-222 while on treatment. | 6 months
  Decreased expression of miRNA-222, has been found during the adipogenic programming of both immortalized and primary hMSCs, suggesting that it acts as negative regulators of fat cell differentiation. We will measure this in plasma.
Changes in glucose and insulin from baseline. | 6 months
  We will measure changes in serum glucose and insulin from baseline while on treatment using ELISA (enzyme-linked immunosorbent assay).
Changes in systolic blood pressure. | 6 months
  We will measure systolic blood pressure changes from baseline while on treatment.
Changes diastolic blood pressure. | 6 months
  We will measure diastolic blood pressure changes from baseline while on treatment.
Changes in heart rate. | 6 months
  We will measure heart rate changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios K. Dimitriadis, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (1):
- WISDEM Centre, University Hospitals Coventry and Warwickshire, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James WP. WHO recognition of the global obesity epidemic. Int J Obes (Lond). 2008 Dec;32 Suppl 7:S120-6. doi: 10.1038/ijo.2008.247. PMID 19136980
- [Background] WHO annual report 2017; Obesity update - © OECD 2017
- [Background] http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/2010/ucm198638.htm
- [Background] FDA approves weight-management drug Saxenda
- [Background] Daviss, Bennett (April 2005).
- [Background] Jordan KW, Nordenstam J, Lauwers GY, Rothenberger DA, Alavi K, Garwood M, Cheng LL. Metabolomic characterization of human rectal adenocarcinoma with intact tissue magnetic resonance spectroscopy. Dis Colon Rectum. 2009 Mar;52(3):520-5. doi: 10.1007/DCR.0b013e31819c9a2c. PMID 19333056
- [Background] Ambros V. The functions of animal microRNAs. Nature. 2004 Sep 16;431(7006):350-5. doi: 10.1038/nature02871. PMID 15372042
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Extracellular/Circulating MicroRNAs: Release Mechanisms, Functions and Challenges